CLINICAL TRIAL: NCT06090006
Title: An Adolescent Health and Wellbeing Check-up Programme in Three African Cities (Y-Check): Protocol for a Multimethod, Prospective, Hybrid Implementation-effectiveness Study
Brief Title: An Adolescent Health and Wellbeing Check-up Programme in Three African Cities (Y-Check)
Acronym: Y-Check
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: World Health Organization (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other); University of Ghana (Other); Mwanza Intervention Trials Unit (Other); Biomedical Research and Training Institute (Other)
Responsible Party: Principal Investigator, Prerna Banati, Scientist, Principal Investigator, World Health Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: WHO ERC.0003778
Record Dates: First submitted 2023-05-16; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Adolescent Development; Adolescent Behavior; Health-Related Behavior; Health Care Seeking Behavior
MeSH Terms: conditions — Adolescent Behavior; Health Behavior; Patient Acceptance of Health Care | interventions — Diet; Mass Screening; HIV Testing

STUDY DESIGN:
Intervention Model Description: In our study sites, a contemporaneous comparison group is not required since no routine screening is currently taking place, and as a result, assessments at baseline will serve as the counterfactual for internal comparisons
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- No comparison group (Other): In our study sites, a contemporaneous comparison group is not required since no routine screening is currently taking place, and as a result, assessments at baseline will serve as the counterfactual for internal comparisons
  Interventions: Other: Screening package; Diagnostic Test: Psychosocial and mental health disorder screening; Diagnostic Test: Alcohol, tobacco and substance use screening; Behavioral: Diet and physical activity screening; Diagnostic Test: Underweight and overweight screening; Diagnostic Test: Anemia; Behavioral: Oral health screening; Behavioral: Circumcision screening; Behavioral: Risky behaviours; Diagnostic Test: HIV testing; Diagnostic Test: STI (CT, NG, TV) testing; Behavioral: Immunization screening; Diagnostic Test: Visual impairment screening; Diagnostic Test: Hearing screening; Diagnostic Test: Physical impairment screening; Diagnostic Test: Uncontrolled epilepsy screening; Diagnostic Test: Pre-hypertension screening

INTERVENTIONS:
Other: Screening package — Y-Check is a novel intervention delivering a health check-up and where indicated will provide on-the-spot care and referral for common conditions on two occasions in adolescence (in young adolescents (10-14 year-olds) - soon after the onset of puberty - and again in older adolescents (15-19 year-olds) - when many adolescents become, or are soon to become, sexually active). It will also provide health promotion information and materials to support positive behaviours and healthy lifestyles during adolescence and beyond. Adolescents will only be screened for conditions that have an accurate, low-cost, acceptable screening test and a locally accessible, effective intervention. The conditions selected for screening will be chosen to reflect the local epidemiological contexts (e.g. screening for malaria will only take place in high malaria endemic areas).
  Other Names: Check ups
Diagnostic Test: Psychosocial and mental health disorder screening — HEEADSSS stands for Home, Education/Employment, Eating, Activities, Drugs, Sexuality, Suicide/Depression, and Safety (Klein et al., 2014) and Patients´ Health Questionnaire - Adolescent (PHQ-A), Generalised Anxiety Disorder (GAD-9) and counselling and referral where indicated
Diagnostic Test: Alcohol, tobacco and substance use screening — World Health Organization (WHO) ASSIST-Y tool (Humeniuk, 2016) and referral where indicated
Behavioral: Diet and physical activity screening — HEEADSSS (Klein et al., 2014) and counselling and advice
Diagnostic Test: Underweight and overweight screening — MUAC (Middle Upper Arm Circumference), BMI (Body Mass Index) followed by Counselling and advice +/- referral where indicated
Diagnostic Test: Anemia — Hemocue. Iron and folic-acid supplementation (3 months supply) if anaemic. If severely anaemic (<8g/dl) refer to health facility.
Behavioral: Oral health screening — Questions on oral health and visual inspection followed by advice, gift of toothpaste and toothbrush, fluoride varnish application +/- Silver Diamine Fluoride application +/- referral
Behavioral: Circumcision screening — Question on circumcision status. Visual inspection. Referral for Voluntary Medical Male Circumcision) where uncircumcised (males only)
Behavioral: Risky behaviours — Question (s) on sexual activity and other risky behaviours, followed by Risk reduction counselling, Provision of condoms, Provision of modern contraceptives (emergency contraception, depot injections, oral contraceptive pill) (females only) PreExposure Prophylaxis (PrEP) (females only)
Diagnostic Test: HIV testing — HIV oral mucosal self-test +/- confirmatory blood-based rapid diagnostic test followed by Counselling + referral to treatment where indicated
Diagnostic Test: STI (CT, NG, TV) testing — Chlamydia Trachomatic (CT) /Neisseria Gonorrhea (NG) test on urine sample, Trichomoniasis Vaginalis (TV) test and treatment where indicated
Behavioral: Immunization screening — Question on Human Papilloma Virus (HPV) immunisation history. Review of vaccination card. Followed by referral to immunization
Diagnostic Test: Visual impairment screening — Peek Acuity or Snellen Tumbling-E and Refer to specialist if indicated
Diagnostic Test: Hearing screening — HearScreen smartphone app +/- HearTest plus Inspection for presence of wax and wax removal.
  Refer to specialist if indicated
Diagnostic Test: Physical impairment screening — Questions on physical impairment. Jump or squat test Functional reach test Referral to specialist if indicated
Diagnostic Test: Uncontrolled epilepsy screening — Questions on experience of convulsions followed by referral to specialist if indicated
Diagnostic Test: Pre-hypertension screening — Blood pressure measured using digital sphygmomanometer followed by counselling and advice if indicated

SUMMARY:
This is a multi-country prospective intervention study, with a mixed-method process evaluation to assess the implementation, effects and short-term cost-effectiveness of Y-Check. The intervention involves screening, on-the-spot care and, if needed, referral of adolescents through health and wellbeing check-up visits in early adolescence (10-14 years) and older adolescence (15-19 years old). In each city, the intervention will be delivered to 2000 adolescents recruited in schools (both age groups) or community venues (older adolescents only).

DETAILED DESCRIPTION:
Background: During adolescence, behaviours are initiated that will have substantial positive or negative impacts on the individual's short- and long-term health and wellbeing, educational attainment and employment prospects. However, adolescents rarely have regular contact with health services, especially for health promotion and disease prevention, and services are not always appropriate for their needs. The investigators co-developed with adolescents a health and wellbeing check-up programme, to improve adolescent health and wellbeing (Y-Check). This paper describes the methods to evaluate the feasibility, acceptability, short-term effects, and cost-effectiveness of Y-Check in three African cities: Cape Coast in Ghana, Mwanza in Tanzania and Chitungwiza in Zimbabwe.

Method: This is a multi-country prospective intervention study, with a mixed-method process evaluation to assess the implementation, effects and short-term cost-effectiveness of Y-Check. The intervention involves screening, on-the-spot care and, if needed, referral of adolescents through health and wellbeing check-up visits in early adolescence (10-14 years) and older adolescence (15-19 years old). In each city, the intervention will be delivered to 2000 adolescents recruited in schools (both age groups) or community venues (older adolescents only). The adolescents will be followed-up at 4 months (all sites) and 12 months (Zimbabwe only). The study will assess the effects of Y-Check on knowledge and behaviours, as well as clinical outcomes and costs. The primary outcome will be the proportion of those screening positive for at least one condition who receive appropriate on-the-spot care or complete appropriate referral for all identified conditions within four months. Secondary outcomes include yield of untreated conditions, reported health-related risk and protective behaviours, engagement with health services, wellbeing, clinical and educational outcomes. A process evaluation will understand acceptability, feasibility, uptake, and fidelity, and an economic evaluation will explore cost effectiveness.

Discussion: This study is innovative in evaluating a comprehensive adolescent health and wellbeing check-up intervention which addresses both health conditions that impact on wellbeing during adolescence, and risk factors for non-communicable diseases in three African cities. Evidence of the intervention´s feasibility, acceptability, and short-term positive effects and costs will support larger scale intervention implementation and rigorous evaluation.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study, adolescents aged 10-19 must fall into one of the first three categories below and fulfil category 4.

1. Be attending selected classes of Year 5 of primary school in Mwanza (median age 11 years); Grade 5/6 of primary school in Chitungwiza (median age 11 years); or Year 1 of Junior Secondary School in Cape Coast (median age 12 years) OR
2. Be attending selected classes in Year 3 of Secondary School in Mwanza (median age 17 years), Form 3/4 in Chitungwiza (median age 17 years), or Year 2 of Senior Secondary School in Cape Coast (median age 16 years) OR
3. Be resident in a selected community during the time of the Y-Check intervention, and be aged 16-19 years AND
4. Have a completed and signed Informed Consent and have a signed Informed Assent Form if the adolescent is below the national age of consent or is seen in a school, irrespective of their age.

Exclusion Criteria:

Not meeting above inclusion criteria

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — 50% males and 50% females
Enrollment: 6000 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Y-Check Screening outcome | 16 weeks (4 months)
  Proportion of those screening positive for at least one condition who receive appropriate on-the-spot care or complete appropriate referral for all identified conditions within 4 months (i.e. they attend a provider for referral care who has been accredited by the study team and has been shown to be capable of providing appropriate referral care).

SECONDARY OUTCOMES:
Condition Screening outcome | 16 weeks (4 months)
  Proportion of those screening positive for each condition who receive appropriate on-the-spot care or complete appropriate referral for that condition within 4 months.
Previously untreated conditions identified (yield) | 16 weeks (4 months)
  This will be measured as: Numerator: number of individuals identified with a condition that is not currently being treated and requires counselling and/or treatment
  Denominator: number of individuals who were screened for the condition.
Qualitative assessment of adolescents who find the intervention acceptable | 16 weeks (4 months)
  Qualitative assessment tool for acceptability of adolescent wellbeing interventions
Qualitative assessment of teachers, parents and health workers who find the intervention acceptable | 16 weeks (4 months)
  Qualitative assessment tool for acceptability of adolescent wellbeing interventions
Proportion of adolescents who take up and use Y-Check services and referrals | 16 weeks (4 months)
  Proportion of young people invited who complete the screening program; proportion of young people invited who complete referrals. Qualitative assessment tool will also be used to assess intervention adoption
Qualitative assessment of perceived value of the intervention to adolescents and to other stakeholders. | 16 weeks (4 months)
  Intervention appropriateness (perceived fit, perceived relevance, perceived usefulness): perceived value of the intervention to adolescents and to other stakeholders.
Proportion of Y-Check visits completed | 16 weeks (4 months)
  Intervention feasibility (actual fit, practicability): Y-Check visits completed
Proportion of referrals completed | 16 weeks (4 months)
  Intervention feasibility (actual fit, practicability): Referrals completed
Proportion of youth reporting youth friendly health services received with quality | 16 weeks (4 months)
  youth-friendly health services quality assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Prerna Banati, PhD, Principal Investigator — World Health Organization; Baltag Valentina, MD, Principal Investigator — World Health Organization; Aoife Doyl, PhD, Principal Investigator — Biomedical Training and Research Institute; Saidi Kapiga, MD, Principal Investigator — Mwanza Intervention Trials Unit; Benedict Weobong, PhD, Principal Investigator — University of Ghana
Locations (3):
- Schools and Community Centers, Cape Coast, Ghana
- Schools and community centers, Mwanza, Tanzania
- Schools and community centers, Chitungwiza, Zimbabwe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banati P, Ross DA, Weobong B, Kapiga S, Weiss HA, Baltag V, Nzvere F, Glozah F, Nsanya MK, Greco G, Ferrand R, Doyle AM; Y-Check Research Programme Team. Adolescent health and well-being check-up programme in three African cities (Y-Check): protocol for a multimethod, prospective, hybrid implementation-effectiveness study. BMJ Open. 2024 Jun 21;14(6):e077533. doi: 10.1136/bmjopen-2023-077533. PMID 38908843
- See also: Summary of Y-Check Phase 2 — https://www.who.int/publications/m/item/ycheck-phase-2-the-effectiveness-and-cost-effectiveness-of-adolescent-health-and-well-being-in-three-african-cities